CLINICAL TRIAL: NCT03075397
Title: VIH-1 Colo-rectal Transmission by Infected Semen Cells and Effects of Seminal Plasma ex Vivo
Brief Title: VIH-1 Colo-rectal Transmission by Infected Semen Cells and Effects of Seminal Plasma ex Vivo (CellspermVIH)
Acronym: CellspermVIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/16/8193; 2016-A01025-46 (Other: ID-RCB)
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection
Keywords: HIV-1; Colo-rectal transmission; seminal plasma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV-1 infected patients (Other): Blood sample and sperm sample are collected
  Interventions: Other: blood sample; Other: sperm sample

INTERVENTIONS:
Other: blood sample — A sample of HIV-1 infected patients's blood is collected
Other: sperm sample — A sample of HIV-1 infected patients's sperm is collected

SUMMARY:
The objective of our project is to determine the infected seminal cell types and the molecular mechanisms involved in HIV cell-associated transmission in the colo-rectal mucosa, using conditions as close as possible to real life, i.e. seminal leukocytes and seminal plasma from HIV-infected donors and tissue explants

DETAILED DESCRIPTION:
This project relies on:

* our expertise of HIV in semen and male genital tract and our experience in organotypic cultures;
* a network of infectious diseases and reproductive biology clinicians to collect, analyze and process seminal cells and seminal plasma from HIV+ donors;
* the expertise in confocal microscopy and ex vivo colo-rectal model. State of the art culture of colo-rectal tissues, primary cell culture and infection, confocal microscopy, flow cytometry, Polymerase Chain Reaction and Luminex assays for cytokine measurements will be the methodologies primarily used in this project.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients who have never been treated by antiretroviral therapy
* Signature of informed consent
* Affiliation to social service

Exclusion Criteria:

* Patients' general condition not allowing protocol follow-up
* Patients with an ejaculation disorder
* Patients unable to perform semen sampling
* Patients with chemotherapy or radiotherapy antecedents
* Patients with very severe oligospermia (≤1million/mL of spermatozoa)
* Patients with active genital infection
* Protected subjects

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Characterize seminal HIV infected cells. | 1 years
  Macrophages and CD4+ T lymphocytes characterization.
Evaluate the potential of seminal HIV infected cells migration and adhesion. | 1 years
  Assess the potential of seminal macrophages and CD4 T cells to adhere and transmigrate.
Determine the efficiency of seminal cell associated infection. | 1 years
  The efficiency of seminal cell associated infection will be determinated in the colo-rectal explants.

SECONDARY OUTCOMES:
Identify molecules expressed and involved in seminal cell adhesion and transmigration. | 1 years
  Identify key adhesion molecules expressed by seminal leucocytes and epithelial cells involved in seminal cell adhesion/transmigration.
Identify seminal and mucosal molecules mediating seminal cell translocation. | 1 years
  Seminal and mucosal soluble molecules mediating seminal cell translocation will be characterized (passive diffusion or active transmigration).
Determine the impact of seminal plasma/cells exposure on mucosal immune cell. | 1 years
  Mucosal immune cell activation, trafficking and the factors involved, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Dejucq-Rainsford, PhD, Study Director — IRSET
Locations (3):
- France (3):
  - CECOS Bretagne Rennes, Rennes, Brittany Region
  - CECOS Hôpital Paule de Viguier, Toulouse, Midi-Pyrénées
  - CECOS Paris Bichat, Paris

IPD SHARING:
Plan to Share IPD: Yes
The duplicated part of the CRFs will then be sent to Mrs DEJUC at the IRST in Rennes, the remaining part will be kept in the investigating center.
  All the data of the study transcribed by the investigator in the CRFs will be transmitted electronically to the person in charge of the data of the INSERM / IRSET 1085 unit. Upon receipt, the data will be entered simply by typing and re-reading on the Excel spreadsheet. The files will be locked by password and backed up daily with storage for 3 months on the server of the INSERM 1085 unit managed by the IT department of the University of Rennes 1. The set Data is saved every evening, with storage for 4 weeks, then archived monthly on tape.

REFERENCES:
- [Background] Roulet V, Satie AP, Ruffault A, Le Tortorec A, Denis H, Guist'hau O, Patard JJ, Rioux-Leclerq N, Gicquel J, Jegou B, Dejucq-Rainsford N. Susceptibility of human testis to human immunodeficiency virus-1 infection in situ and in vitro. Am J Pathol. 2006 Dec;169(6):2094-103. doi: 10.2353/ajpath.2006.060191. PMID 17148672
- [Background] Le Tortorec A, Le Grand R, Denis H, Satie AP, Mannioui K, Roques P, Maillard A, Daniels S, Jegou B, Dejucq-Rainsford N. Infection of semen-producing organs by SIV during the acute and chronic stages of the disease. PLoS One. 2008 Mar 12;3(3):e1792. doi: 10.1371/journal.pone.0001792. PMID 18347738
- [Background] Le Tortorec A, Satie AP, Denis H, Rioux-Leclercq N, Havard L, Ruffault A, Jegou B, Dejucq-Rainsford N. Human prostate supports more efficient replication of HIV-1 R5 than X4 strains ex vivo. Retrovirology. 2008 Dec 31;5:119. doi: 10.1186/1742-4690-5-119. PMID 19117522
- [Background] Houzet L, Matusali G, Dejucq-Rainsford N. Origins of HIV-infected leukocytes and virions in semen. J Infect Dis. 2014 Dec 15;210 Suppl 3:S622-30. doi: 10.1093/infdis/jiu328. PMID 25414416
- [Background] Camus C, Matusali G, Bourry O, Mahe D, Aubry F, Bujan L, Pasquier C, Massip P, Ravel C, Zirafi O, Munch J, Roan NR, Pineau C, Dejucq-Rainsford N. Comparison of the effect of semen from HIV-infected and uninfected men on CD4+ T-cell infection. AIDS. 2016 May 15;30(8):1197-208. doi: 10.1097/QAD.0000000000001048. PMID 26854806
- [Background] Anderson DJ, Politch JA, Nadolski AM, Blaskewicz CD, Pudney J, Mayer KH. Targeting Trojan Horse leukocytes for HIV prevention. AIDS. 2010 Jan 16;24(2):163-87. doi: 10.1097/QAD.0b013e32833424c8. No abstract available. PMID 20010071